CLINICAL TRIAL: NCT04461821
Title: Exhaled Breath Analysis by Secondary Electrospray Ionization - Mass Spectrometry in Children and Adolescents (EBECA)
Brief Title: Exhaled Breath Analysis by Secondary Electrospray Ionization - Mass Spectrometry in Children and Adolescents
Acronym: EBECA
Status: Recruiting | Type: Observational
Sponsor: University Children's Hospital Basel (Other)
Collaborators: Swiss National Science Foundation (Other); Fondation Botnar (Switzerland) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2020-00778; ks20Sinues
Record Dates: First submitted 2020-06-23; First posted 2020-07-08 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Respiratory Diseases; Neurological Disorders; Type 1 Diabetes
Keywords: Exhaled breath analysis; Therapeutic drug monitoring (TDM); Secondary Electrospray ionization - mass spectrometry (SESI-MS); breath analysis platform; breath metabolomics
MeSH Terms: conditions — Respiratory Tract Diseases; Nervous System Diseases; Diabetes Mellitus, Type 1 | interventions — Hematologic Tests; Urinalysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be divided into two sets and stored at -80°C in a dedicated, lock-secured laboratory freezer for later molecular analysis. One set will be used for blood plasma metabolomics. A second set will be analyzed depending on the exploratory findings regarding breath compounds. These samples shall enable retrospective correlation between the concentrations of molecules-of-interest in breath and blood.
  Saliva and urine samples will be divided in two sets and stored at -80°C in a dedicated, lock-secured laboratory freezer for later molecular analysis. One set will be used for metabolomics. A second set will be analyzed depending on the exploratory findings regarding breath compounds. These samples shall enable retrospective correlation between the concentrations of molecules-of-interest in breath and saliva.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (12):
- obstructive bronchitis/bronchiolitis
  Interventions: Diagnostic Test: Real-time SESI-MS breath analysis; Diagnostic Test: Off-line breath analysis; Diagnostic Test: Blood analysis
- pneumonia
  Interventions: Diagnostic Test: Real-time SESI-MS breath analysis; Diagnostic Test: Off-line breath analysis; Diagnostic Test: Blood analysis
- asthma
  Interventions: Diagnostic Test: Real-time SESI-MS breath analysis; Diagnostic Test: Off-line breath analysis; Diagnostic Test: Blood analysis
- neurological diseases
  Interventions: Diagnostic Test: Real-time SESI-MS breath analysis; Diagnostic Test: Off-line breath analysis; Diagnostic Test: Blood analysis
- type 1 diabetes (T1D)
  Interventions: Diagnostic Test: Real-time SESI-MS breath analysis; Diagnostic Test: Off-line breath analysis; Diagnostic Test: Blood analysis; Diagnostic Test: Saliva analysis; Diagnostic Test: Urine analysis
- pharmacotherapy with bronchodilators
  Interventions: Diagnostic Test: Real-time SESI-MS breath analysis; Diagnostic Test: Off-line breath analysis; Diagnostic Test: Blood analysis
- pharmacotherapy with antibiotics
  Interventions: Diagnostic Test: Real-time SESI-MS breath analysis; Diagnostic Test: Off-line breath analysis; Diagnostic Test: Blood analysis
- pharmacotherapy with antiviral medication
  Interventions: Diagnostic Test: Real-time SESI-MS breath analysis; Diagnostic Test: Off-line breath analysis; Diagnostic Test: Blood analysis
- pharmacotherapy with antifungal medication
  Interventions: Diagnostic Test: Real-time SESI-MS breath analysis; Diagnostic Test: Off-line breath analysis; Diagnostic Test: Blood analysis
- pharmacotherapy with antiepileptic medication
  Interventions: Diagnostic Test: Real-time SESI-MS breath analysis; Diagnostic Test: Off-line breath analysis; Diagnostic Test: Blood analysis
- pharmacotherapy with immuno suppressants and immune-modulati
  Interventions: Diagnostic Test: Real-time SESI-MS breath analysis; Diagnostic Test: Off-line breath analysis; Diagnostic Test: Blood analysis
- pharmacotherapy with anesthesia (including sedating, analges
  Interventions: Diagnostic Test: Real-time SESI-MS breath analysis; Diagnostic Test: Off-line breath analysis; Diagnostic Test: Blood analysis

INTERVENTIONS:
Diagnostic Test: Real-time SESI-MS breath analysis — Participants will be asked to refrain from eating, drinking, chewing gum use or brushing their teeth at least 1 hour before the measurements will be performed. Room temperature and lighting will be set at the same level for all measurements. Participants will exhale through a disposable mouthpiece into a commercially available SESI source (FIT S.L., Spain). While performing full exhalations, the subjects will keep the pressure through the sampling line at a fixed value monitored by a digital manometer. Breath prints will be collected in real-time recording multiple replicates (typically six in positive and negative ion mode). The whole procedure is absolutely non-invasive and is usually accomplished without any effort in around 15 min per subject.
Diagnostic Test: Off-line breath analysis — In young children below the age of 4 not capable of completing the on-line exhalation maneuvers, or in cases when the patient needs cannot approach the mass spectrometer, the sample will be collected off-line. They will be asked to exhale into a bag that will be transported to the lab and deflated into the mass spectrometer for analysis. Exhaled breath of patients under anesthesia will also collected using available ventilation system in the operation theatre.
Diagnostic Test: Blood analysis — Blood analysis done in patients who undergo regular blood sampling needed for clinical routine laboratory controls. This includes i) children and adolescents receiving medications which require TDM ii) patients with acute diseases such as TD1 and pneumonia and iii) patients with chronic diseases such as asthma bronchiale. For those patients where a blood sample is drawn during the clinical routine, an additional blood sample consisting of only several blood drops will be collected using the same blood sampling line. No additional venous puncture for research purpose will be done.
Diagnostic Test: Saliva analysis — During the diagnostic and therapeutic work-up of T1D patients, saliva samples are collected during the clinical routine. For those patients, additional samples will be obtained by clinically trained investigators.
  Groups: type 1 diabetes (T1D)
Diagnostic Test: Urine analysis — During the diagnostic and therapeutic work-up of T1D patients, urine samples are collected during the clinical routine. For those patients, additional samples will be obtained by clinically trained investigators.
  Groups: type 1 diabetes (T1D)

SUMMARY:
This study is to investigate breath analysis (breath metabolomics) combined with established bioinformatic tools as a platform for companion diagnostics.

DETAILED DESCRIPTION:
Therapeutic drug monitoring (TDM) is defined as measuring concentrations of a drug at one or more time points in a biological matrix after a dose. The purpose of TDM is to individualize the drug dose to achieve maximum efficacy and at the same time minimize toxicity. The concept of TDM could potentially be even more valuable if in addition to drug concentrations, other drug-regulated and drug-related metabolites could be included in the models to define optimal dosage. There exists a clinical need to stratify patients with better precision to improve current clinical and therapeutic management. Breath analysis offers an opportunity to non-invasively retrieve relevant information on the ongoing internal biochemical processes, as well as to monitor the respiratory system itself. For breath analysis, a Secondary Electrospray ionization - mass spectrometry (SESI-MS) breath analysis platform will be used to capture disease-related, drug-regulated and drug-related metabolites (breath metabolomics) in exhaled breath. This information, retrieved in parallel to standard of care clinical co-variates, could have the potential to provide a more personalized therapeutic management of patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 0 ≤ 22 years at study entry and signed informed consent

Additional inclusion criteria for respiratory disease population:

* Acute disease: - Acute signs for a respiratory disease, indicated by e.g. increased work of breathing (e.g. dyspnea, increased respiratory rate), cough or wheezing.
* Chronic disease: - Suspected or confirmed chronic airway disease (e.g. asthma).

Additional inclusion criteria for neurological disease population:

* Acute disease: - Acute presentation or report within 24 hours of any signs of neurological deficit (motor function, sensoneural, or verbal).
* Chronic disease: - Confirmed chronic neurologic disease (e.g. childhood epilepsy).

Additional inclusion criteria for T1D disease population:

* Acute disease: - Hyperglycemia and/or pH (venous) <7.3, bicarbonate >10 mmol/L, increased levels of acetone in blood or urine in the context of newly diagnosed or known T1D.
* Chronic disease: - Confirmed diagnosis of T1D

Exclusion Criteria:

* Physical or intellectual impairment precluding protocol adherence.

Additional exclusion criteria for respiratory disease population:

* Known malignancy, active smoker (passive smoke exposure is not an exclusion criterium), known inflammatory diseases (e.g. autoimmune disease) that require medical and/or pharmacological treatment and is associated with an inflammatory response, relevant congenital defects

Additional exclusion criteria for neurological disease population:

* Known malignancy, active smoker (passive smoke exposure is not an exclusion criterium), known inflammatory diseases (e.g. autoimmune disease) that require medical and/or pharmacological treatment and is associated with an inflammatory response, relevant congenital defects.

Additional exclusion criteria for T1D population:

* Known malignancy, active smoker (passive smoke exposure is not an exclusion criterium), relevant congenital defects.

Max Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants presenting with an acute disease in the emergency department at the University of Basel Children's Hospital (UKBB).
  Participants with chronic diseases recorded at the University of Basel Children's Hospital (UKBB).
Sampling Method: Probability Sample
Enrollment: 3600 (Estimated)
Dates: Start 2020-09-11 (Actual); Primary Completion 2030-07 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Days of hospitalization | approx 30 days (from beginn hospitalisation to discharge date)
  In the presentation of an acute disease the primary outcome will be days of hospitalization and its association with the exhaled breath pattern.
Change in Mass spectrometric profile of exhaled breath patterns | Week 0 (first regular clinic visit) to Follow-up visits (approx. years 1-10)
  In the chronic presentation of the diseases, the mass spectrometric profile of exhaled breath patterns is analyzed
Change in Concentration of exhaled metabolites of pharmacotherapy | Week 0 (first regular clinic visit) to Follow-up visits (approx. years 1-10)
  Concentration of exhaled metabolites of pharmacotherapy (breath metabolomics data)

SECONDARY OUTCOMES:
Identification of chemical structure of exhaled molecules (acetone, glucose) | approx 30 days (from begin hospitalisation to discharge date)
  Identification of chemical structure of exhaled molecules (acetone, glucose)
Correlations of identified molecules (acetone, glucose) in exhaled breath with body fluids (blood, saliva, urine) for T1D acute disease (mmol/l) | 0h, 2h, 4h, 6h, 8h, 12h, 18h, 24h, 36h, 48h, 72h (h =hours after hospital admission)
  Correlations of identified molecules (acetone, glucose) in exhaled breath with body fluids (blood, saliva, urine) for T1D acute disease (mmol/l)
Change in clinical endpoint lung function (Forced Expiratory Pressure in 1 Second FEV1 l/s) for correlation between clinical endpoint and the abundance of exhaled metabolites | approx 10 years (from begin hospitalisation to discharge date and from first regular clinic visit to Follow-up visits)
  Change in clinical endpoint lung function (Forced Expiratory Pressure in 1 Second FEV1 l/s) for correlation between clinical endpoint and the abundance of exhaled metabolites
Change in clinical endpoint (body temperature, Celsius) for correlation between clinical endpoint and the abundance of exhaled metabolites | approx 10 years (from begin hospitalisation to discharge date and from first regular clinic visit to Follow-up visits)
  Change in clinical endpoint (body temperature) for correlation between clinical endpoint and the abundance of exhaled metabolites
Change in clinical endpoint (blood pressure, mmHg) for correlation between clinical endpoint and the abundance of exhaled metabolites | approx 10 years (from begin hospitalisation to discharge date and from first regular clinic visit to Follow-up visits)
  Change in clinical endpoint (blood pressure) for correlation between clinical endpoint and the abundance of exhaled metabolites

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Sinues, Prof. Dr., Principal Investigator — University Children's Hospital Basel, UKBB
Locations (1):
- University Children's Hospital Basel (UKBB), Basel, Switzerland

REFERENCES:
- [Derived] Zeng J, Stankovic N, Singh KD, Steiner R, Frey U, Erb T, Sinues P. Breath Analysis of Propofol and Associated Metabolic Signatures: A Pilot Study Using Secondary Electrospray Ionization-High-resolution Mass Spectrometry. Anesthesiology. 2025 Aug 1;143(2):345-356. doi: 10.1097/ALN.0000000000005531. Epub 2025 Apr 21. PMID 40258137